CLINICAL TRIAL: NCT01621477
Title: T-Cell Replete Haploidentical Donor Hematopoietic Stem Cell Plus Natural Killer (NK) Cell Transplantation in Patients With Hematologic Malignancies Relapsed or Refractory Despite Previous Allogeneic Transplant
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated in August 2016 due to replacement by a new study.
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Assisi Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HAP3R; NCI-2012-00554 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2012-06-08; First posted 2012-06-18 (Estimated); Results first posted 2017-02-20 (Actual); Last update posted 2017-02-20 (Actual); Status verified 2016-12

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myelocytic Leukemia; Chronic Myelocytic Leukemia; Juvenile Myelomonocytic Leukemia; Myelodysplastic Syndrome; Hodgkin or Non-Hodgkin Lymphoma; Sarcoma, Myeloid
Keywords: Hematologic malignancy; Hematopoietic cell transplant
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myelomonocytic, Juvenile; Myelodysplastic Syndromes; Lymphoma, Non-Hodgkin; Sarcoma, Myeloid; Hematologic Neoplasms | interventions — Clofarabine; Cytarabine; Busulfan; plerixafor; Cyclophosphamide; thymoglobulin; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): All study participants.
  Interventions: clofarabine, cytarabine, busulfan, plerixafor, cyclophosphamide, antithymocyte globulin (rabbit), stem cells, tacrolimus, mycophenolate mofetil
  Interventions: Drug: clofarabine; Drug: cytarabine; Drug: busulfan; Drug: Plerixafor; Drug: cyclophosphamide; Drug: antithymocyte globulin (rabbit); Biological: stem cells; Drug: Tacrolimus; Drug: mycophenolate mofetil

INTERVENTIONS:
Drug: clofarabine — Given on Day -9 and Day -8 (Day 0 is first stem cell infusion). Drug class: antineoplastic agent
  Other Names: Cl-F-Ara-A; CAFdA; Clofarex; Clolar(TM)
Drug: cytarabine — Given on Day -9 and Day -8 (Day 0 is first stem cell infusion). Drug class: antineoplastic agent
  Other Names: Ara-C
Drug: busulfan — Given on Day -7 and Day -6 (Day 0 is first stem cell infusion). Drug class: antineoplastic agent
  Other Names: Myleran(R); Busulfex
Drug: Plerixafor — Given on Day -7 and Day -6 (Day 0 is first stem cell infusion). Drug class: Hematopoietic Stem Cell Mobilizer
  Other Names: AMD3100; Mozobil(R)
Drug: cyclophosphamide — Given on Day -5 and Day +4 (Day 0 is first stem cell infusion). Drug class: antineoplastic agent; immunosuppressive agent.
  Other Names: Cytoxan
Drug: antithymocyte globulin (rabbit) — Given on Day -4, Day -3, Day -2, and Day -1 (Day 0 is first stem cell infusion). Drug class: immunosuppressive agent.
  Other Names: Rabbit ATG; Rabbit Thymoglobulin(R)
Biological: stem cells — Patients undergo T cell replete Hematopoietic stem cell infusion on Day 0 and Day +1. Patients undergo natural killer (NK) cell transplantation on day +6 (Day 0 is first stem cell infusion).
  Other Names: HSC infusion
Drug: Tacrolimus — Given on Day +11 (Day 0 is first stem cell infusion). Drug class: immunosuppressive agent.
  Other Names: FK506; Prograf(R); Protonic(R)
Drug: mycophenolate mofetil — Given on Day +11 (Day 0 is first stem cell infusion). Drug class: immunosuppressive agent.
  Other Names: MMF; CellCept(R)

SUMMARY:
The primary aim of this protocol is to evaluate if the one-year survival is significantly improved in the group of patients who receive a T-cell replete haploidentical donor hematopoietic cell transplant (HCT) with a novel reduced intensity conditioning regimen. Study population will consist of patients (21 years or under) with hematologic malignancies that have relapsed or are refractory after prior allogeneic transplant. Toxicity will be evaluated by the rate of transplant related mortality and the rates of moderate and severe graft-versus-host disease (GvHD) at day 100. The investigators will describe event-free, and disease-free survival at one year, as well as the rates of hematopoietic recovery and donor engraftment and study comprehensively immune reconstitution following T-cell replete haploidentical transplantation.

DETAILED DESCRIPTION:
Patients with refractory hematologic malignancies, including those who develop recurrent disease after allogeneic hematopoietic cell transplantation, have a dismal prognosis. Historically, both regimen-related mortality and disease recurrence have been significant causes of treatment failure in this heavily pre-treated patient population. Our institution has utilized mismatched family member (haploidentical) donors for these patients for a number of years for the following reasons: (1) Only 30% of patients have matched related donors available; (2) transplantation can be performed more rapidly since the time to unrelated donor transplantation averages 3 to 4 months; (3) no other curative treatment options are available. These therapeutic interventions have been largely successful given the dismal prognosis in this patient group; however disease recurrence remains the most significant cause of treatment failure. To provide maximum benefit for this challenging population, the goals of a therapeutic transplant protocol should include: (1) a conditioning regimen that is well tolerated, even in a heavily pre-treated population; but it should also provide substantial antileukemia effects, and (2) should establish rapid immune recovery such that the patient may benefit from graft versus leukemia effect and early protection from life threatening infections while also limiting dangerous and counter-productive graft versus host disease.

The primary aim of this protocol will be to evaluate if the one-year survival is significantly improved in the group of patients receiving T-cell replete haploidentical donor HCT with a novel clofarabine, cytarabine, busulfan, plerixafor, cyclophosphamide, and ATG based reduced intensity conditioning regimen whose hematologic malignancy has relapsed or is refractory after prior allogeneic transplant. Toxicity will be evaluated by the rate of transplant related mortality and the rates of moderate and severe graft versus host disease at day 100. The investigators will also describe event-free, and disease-free survival at one year, as well as the rates of hematopoietic recovery and donor engraftment. Additionally, the investigators will study comprehensively immune reconstitution following T-cell replete haploidentical transplantation.

PRIMARY OBJECTIVE:

* Evaluate if the one-year survival is significantly improved in a group of children receiving a therapeutic regimen for high-risk hematologic malignancy that is relapsed or refractory despite previous allogeneic hematopoietic cell transplantation (HCT) using a novel reduced intensity conditioning and T-cell replete haploidentical donor hematopoietic stem cell plus NK cell transplantation.

SECONDARY OBJECTIVES:

* Estimate the incidence of malignant relapse, event-free survival, and disease free survival (DFS) at one-year post-transplantation.
* Estimate incidence and severity of acute and chronic (GVHD).
* Estimate the rate of transplant related mortality (TRM) in the first 100 days after transplantation.

ELIGIBILITY:
Inclusion Criteria - for transplant recipient:

* Age less than 21 years.
* One of the following hematologic malignancies that has relapsed or remains refractory after prior allogeneic HCT:

  * Acute lymphoblastic leukemia (ALL)
  * Acute myeloid leukemia (AML) (including myeloid sarcoma)
  * Chronic myelogenous leukemia (CML), juvenile myelomonocytic leukemia (JMML), myelodysplastic syndrome (MDS), Hodgkin or non-Hodgkin lymphoma (NHL)
* Has a suitable single haplotype matched (≥ 3 of 6) family member donor.
* Does not have any other active malignancy other than the one for which this transplant is indicated.
* If prior central nervous system (CNS) leukemia, it must be treated and have no evidence of CNS disease
* Does not have current uncontrolled bacterial, fungal, or viral infection per the judgment of the principal investigator.
* Patient must fulfill pre-transplant evaluation:

  * Left ventricular ejection fraction greater than 40%, or shortening fraction greater than or equal to 25%.
  * Creatinine clearance or Glomerular Filtration Rate of ≥70 ml/min/1.73m^2.
  * Forced vital capacity (FVC) ≥ 40% of predicted value; or pulse oximetry ≥ 92% on room air if patient is unable to perform pulmonary function testing.
  * Karnofsky or Lansky (age-dependent) performance score ≥ 50.
  * Total bilirubin ≤ 1.5 times the upper limit of normal for age.
  * Alanine aminotransferase (ALT) ≤ 3 times the upper limit of normal for age.
  * Not pregnant. If female with child bearing potential, must be confirmed by negative serum or urine pregnancy test within 14 days prior to enrollment.
  * Not breast feeding.
  * Does not have active acute bronchiolitis obliterans or bronchiolitis obliterans organizing pneumonia.

Inclusion Criteria - for donor:

* At least single haplotype matched (≥ 3 of 6) family member,
* At least 18 years of age.
* Human immunodeficiency virus (HIV) negative.
* Not pregnant as confirmed by negative serum or urine pregnancy test within 14 days prior to enrollment (if female).
* Not breast feeding.
* A suitable donor is identified as either:

  * Has completed the process of donor eligibility determination as outlined in 21 CFR 1271 and agency guidance; OR
  * Does not meet 21 CFR 1271 eligibility requirements, but has a declaration of urgent medical need completed by the principal investigator or physician sub-investigator per 21 CFR 1271.

Exclusion Criteria:

* Does not meet above inclusion criteria.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2012-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brandon M. Triplett, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty four participants were enrolled at St. Jude Children's Research Hospital between August 2012 and November 2014.
Pre-assignment Details: Of the 34 participants enrolled on the study, 17 were donors. Donors did not receive treatment and are not followed for data collection to answer the study objectives. They are therefore not included in the results reported here.
Groups:
- Treatment: Study participants (excluding donors) who were enrolled and underwent transplant.
Period: Overall Study
Arm/Group | Treatment
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment: Study participants (excluding donors) who were enrolled and underwent transplant. Donors did not receive treatment and are not followed for data collection to answer the study objectives. They are therefore not included in the results reported here.
Arm/Group | Treatment
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.84 (5.84)
Age, Continuous [Median (Full Range); unit: years] | 6.97 [0.89 to 19.68]
Gender [Count of Participants; unit: Participants]
  Female | 9
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: One-year Survival (OS)
Description: Evaluate the number of participants alive at 1 year. The number of participants surviving to one-year post-transplantation is given.
Time Frame: One year post transplant
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 17
participants | 7

2. Secondary Outcome: Incidence of Malignant Relapse
Description: Estimate the incidence of malignant relapse at one year post-transplant. The number of participants with malignant relapse or progressive disease is given. Relapse was evaluated using standard WHO criteria for each disease.
Time Frame: One year post transplantation.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 17
participants | 10

3. Secondary Outcome: Event-Free Survival (EFS)
Description: Estimate the EFS at one-year post-transplantation. The event is defined as relapse or death due to any cause. The number of participants who were alive without relapse at one year post-transplant is reported.
Time Frame: one year post transplant
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 17
participants | 4

4. Secondary Outcome: Disease-Free Survival (DFS)
Description: Estimate the DFS at one-year post-transplantation. The event is defined as relapse or death due to relapse. The number of participants who did not relapse up to one year post transplant is reported.
Time Frame: one year post transplant
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 17
participants | 7

5. Secondary Outcome: Incidence and Severity of Acute Graft Versus Host Disease (GVHD)
Description: The number of participants with acute GVHD is given, organized by grade. Participants are graded on a scale from 1 to 4, with 1 being mild and 4 being severe.
Time Frame: 100 days post transplant
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 17
participants
  No Acute GVHD | 9
  Grade I | 3
  Grade II | 1
  Grade III | 3
  Grade IV | 1

6. Secondary Outcome: Incidence and Severity of Chronic Graft Versus Host Disease (GVHD)
Description: The severity of chronic GVHD will be described. Chronic GVHD was evaluated using NIH Consensus Global Severity Scoring. The number of participants with chronic GVHD is given, organized by severity.
Time Frame: 100 days post transplant
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 17
participants
  No Chronic GVHD | 15
  Mild | 0
  Moderate | 2
  Severe | 0

7. Secondary Outcome: Number of Participants With Transplant Related Mortality (TRM)
Description: The number of participants who died due to TRM in the first 100 days post-transplant is given.
Time Frame: 100 days post transplant
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 17
participants | 2

ADVERSE EVENTS:
Time Frame: Participants were followed for adverse events from the start of conditioning therapy and throughout the first year post hematopoietic cell transplant (HCT).
Groups:
- Treatment: Study participants (excluding donors) who were enrolled to receive treatment with clofarabine, cytarabine, busulfan, plerixafor, cyclophosphamide, antithymocyte globulin (rabbit), stem cells, tacrolimus, and mycophenolate mofetil. Donors did not receive treatment and are not followed for data collection to answer the study objectives. They are therefore not included in the results reported here.
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 10/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=17)
Allergic reaction, dexmedetomidine (precedex) (Immune system disorders) | 1 (1)
Graft failure (Blood and lymphatic system disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Thrombotic microangiopathy (disorder) (Blood and lymphatic system disorders) | 1 (1)
Fever without neutropenia (General disorders) | 5 (6)
Stomatitis, viral (Gastrointestinal disorders) | 1 (1)
Hemorrhage, pulmonary (Blood and lymphatic system disorders) | 3 (3)
Hepatitis (Hepatobiliary disorders) | 1 (1)
Febrile neutropenia (Infections and infestations) | 1 (1)
Infection, enterobacter cloacae, blood (Infections and infestations) | 1 (1)
Infection, pseudomonas aeruginosa, disseminated (Infections and infestations) | 1 (1)
Infection, staphylococcus epidermidis, blood (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Apnea (Nervous system disorders) | 1 (1)
Mood alteration (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Subdural hygroma (Nervous system disorders) | 1 (1)
Uremic encephalopathy (disorder) (Nervous system disorders) | 1 (1)
Adult respiratory distress syndrome (disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Interstitial pneumonitis syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nodule, pulmonary lobe of lung, right (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (disorder) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tension pneumothorax, lung, right (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Failure, renal (Renal and urinary disorders) | 1 (1)
Acute infusion reaction, stem cells (General disorders) | 2 (2)
Engraftment syndrome (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=17)
Allergic drug reaction, cefepime (Immune system disorders) | 1 (1)
Allergic drug reaction, vancomycin (Immune system disorders) | 2 (2)
Bradycardia (finding) (Cardiac disorders) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1)
Heart failure (disorder) (Cardiac disorders) | 1 (1)
Hypertension (Cardiac disorders) | 6 (7)
Hypotension (Cardiac disorders) | 3 (4)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pulmonary hypertension (Cardiac disorders) | 2 (2)
Fever without neutropenia (General disorders) | 4 (4)
Neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (1)
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 (1)
Hemorrhagic cystitis (Blood and lymphatic system disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Colitis (Hepatobiliary disorders) | 1 (1)
Veno-occlusive disease, hepatic (Hepatobiliary disorders) | 2 (2)
Candidiasis, oral (Infections and infestations) | 1 (1)
Encephalitis (Infections and infestations) | 1 (1)
Febrile neutropeenia (Infections and infestations) | 15 (25)
Hepatitis (Infections and infestations) | 1 (1)
Infection, adenovirus, respiratory tract (Infections and infestations) | 1 (1)
Infection, adenovirus, stool (Infections and infestations) | 10 (12)
Infection, BK virus, blood (Infections and infestations) | 5 (5)
Infection, BK virus, urine (Infections and infestations) | 4 (4)
Infection, candida parapsilosis, blood (Infections and infestations) | 1 (1)
Infection, coagulase negative staphylococcus, blood (Infections and infestations) | 1 (1)
Infection, enterococcus faecalis, blood (Infections and infestations) | 1 (1)
Infection, Epstein Barr virus, blood (Infections and infestations) | 2 (2)
Infection, human herpes virus 6, blood (Infections and infestations) | 5 (6)
Infection, klebsiella, blood (Infections and infestations) | 1 (1)
Infection, lactobacillus, urinary tract (Infections and infestations) | 1 (1)
Infection, microbacterium aurum, blood (Infections and infestations) | 1 (1)
Infection, parainfluenza type 4, respiratory tract (Infections and infestations) | 1 (1)
Infection, respiratory syncytial virus, respiratory tract (Infections and infestations) | 1 (1)
Infection, rotavirus, stool (Infections and infestations) | 1 (2)
Infection, staphylococcus epidermidis, blood (Infections and infestations) | 1 (1)
Infection, staphylococcus, urine (Infections and infestations) | 1 (1)
Infection, vancomycin resistant enterococcus faecium, stool (Infections and infestations) | 1 (1)
Infection, vancomycin-resistant enterococcus, blood (Infections and infestations) | 2 (3)
Infection, vancomycin resistant enterococcus, rectum (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Reactivation, Epstein Barr virus (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2)
Hemophagocytic lymphohistiocytosis (disorder) (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (disorder) (Metabolism and nutrition disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Obstructive sleep apnea (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Sensory neuropathy (Nervous system disorders) | 1 (1)
Pain, knee, bilateral (General disorders) | 1 (1)
Pain, shoulder, bilateral (General disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pleural effusion, bilateral (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion, right (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cystitis (Renal and urinary disorders) | 1 (1)
Hemorrhagic cystitis (Renal and urinary disorders) | 5 (5)
Acute infusion reaction, NK cells (General disorders) | 1 (1)
Acute infusion reaction, stem cells (General disorders) | 14 (16)
Cytokine release syndrome, ATG (Immune system disorders) | 12 (12)
Engraftment syndrome (General disorders) | 5 (5)
Occlusive thrombus (morphologic abnormality) (Vascular disorders) | 1 (1)
Thrombus, upper extremity and neck, left (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes